CLINICAL TRIAL: NCT06092359
Title: The Eye in Orbit- Analysis of the Anatomical and Functional Ocular Changes Related to Space Flights: UCF Adaptation.
Brief Title: The Eye in Orbit: UCF Adaption
Status: Completed | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003845
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Spaceflight Associated Neuro-Ocular Syndrome; SANS
Keywords: SANS; Spaceflight Associated Neuro-Ocular Syndrome; Optical Coherence Tomography Angiography; OCTA; Space; Astronaut
MeSH Terms: conditions — spaceflight-induced visual impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to understand the impact of space travel on the eyes. Space flight impacts numerous aspects of ocular anatomy and physiology. Current hypotheses are based on pressure changes within and around the optic nerve. Retinal and choroid blood drainage may be affected by microgravity associated cerebrospinal fluid pressure changes. Recently, a new imaging modality, Optical Coherence Tomography Angiography (OCTA), has been able to reveal micro vascular changes in the retina and choroid. To date, no microgravity ocular imaging tests have been published using OCTA. In this study the researchers aim to describe microgravity circadian choroidal and retinal vasculature using multimodal imaging including OCTA to better understand space associated ocular changes.

ELIGIBILITY:
Inclusion Criteria:

- astronauts in the AX1/Rakia mission, which was scheduled for space flight in late March 2022.

Exclusion Criteria:

* adults unable to consent
* individuals who are not yet adults (infants, children, teenagers) -
* pregnant women
* prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study necessarily had a very specific population. The study only enrolled astronauts in the AX1/Rakia mission, which was scheduled for space flight in late March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
To examine early changes in ocular physiology following exposure to microgravity and asses these changes as risk factor for Spaceflight Associated Neuro-Ocular Syndrome (SANS). | 4 months
Asses early changes in ocular physiology as risk factor for Spaceflight Associated Neuro-Ocular Syndrome (SANS). | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Patel, MD, MSc, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No